CLINICAL TRIAL: NCT06634446
Title: Self-administered COgnitive Personalized Training in Early Psychosis: a Randomized Controlled Trial in Adolescents and Young Adults to Assess Efficacy and Efficiency of an EHealth Application Providing Personalized Cognitive Training
Brief Title: Self-administered COgnitive Personalized Training in Early Psychosis
Acronym: SCOPe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D19-P002; 2019 A00399 48 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-10-03; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: First Episode Psychosis (FEP)
Keywords: First Episode Psychosis (FEP),; schizophrenia; Cognitive Personalized training; adolescents and young adults FEP; personalized cognitive training; Chronic psychosis; Biological Testing; Metabolic Alterations
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): the experimental group will use a mobile application for cognitive training for 3 months.
  Interventions: Device: a mobile application for cognitive training
- comparative control group (Active Comparator): Patients in the control group will use video games with no prominent cognitive involvement
  Interventions: Device: video games

INTERVENTIONS:
Device: a mobile application for cognitive training — Personalized cognitive training (PCT) HappyNeuronwill be delivered via a tablet or mobile application for 24 hours within 12 weeks, with a weekly supervision-call to reinforce their motivation.
  HappyNeuron Pro is a digital therapy tool designed for clinicians to provide engaging cognitive therapy via a web-based platform. It is compatible with PC, Mac, iPad, and Android devices and is available in multiple languages. The tool features exercises from established cognitive remediation programs.
  Functionality: The program offers 22 cognitive exercises targeting seven key functions outlined in the MATRICS framework: Processing Speed, Selective Attention, Reasoning and Working Memory, Verbal Memory, Visual Memory, and Auditory Memory. Exercises are customizable to meet individual patient needs, facilitating personalized cognitive training.
  User Experience: Each session comprises brief, self-administered exercises, with the order and difficulty adjusted by clinicians.
  Other Names: cognitive training; HappyNeuron Pro; Personalized cognitive training
  Arms: Experimental group
Device: video games — Patients in the control group will use video games with no prominent cognitive involvement no prominent cognitive involvement
  Arms: comparative control group

SUMMARY:
The overall objective of SCOPe is to improve early intervention in psychosis by providing an innovative eHealth tool that will enable personalized cognitive training, adapted to the individual's cognitive abilities.

Cognitive remediation improves quality of life and functional outcome in patients with chronic psychosis. It would even be more efficacious in the early phase of psychosis by tackling the negative impact of psychosis on education achievement and employment. However, cognitive dysfunctions are often overlooked in FEP and cognitive remediation is not always accessible. New technologies can provide us with youth-friendly, non-stigmatizing tools, such as self administered, training applications so that all first-line clinical settings or professionals, and in fine all patients, can have access, wherever they live, to personalized cognitive training focusing on impaired functions.

Early psychosis can be associated with inflammation, metabolic deficiency, as well as early structural brain anomalies that reflect brain plasticity abilities and could influence the prognosis and response to cognitive training.

Our background hypothesis is that promoting neuroplasticity by cognitive training could attenuate or reverse early cognitive deficits and improve the overall functional outcome in young patients experiencing FEP and that this effect is modulated by individual brain plasticity abilities.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent and young adults, both genders, aged 16 to 35,
* Seeking help in one of the recruiting centers,
* Newly diagnosed as experiencing an Episode of Psychosis (reaching criteria as described in the Comprehensive Assessment of at Risk Mental States (CAARMS) within the year
* Written informed consent signed (and from one legal guardian for minors).

Exclusion Criteria:

* Severe and unstabilized medical conditions,
* Insufficient level in reading and/or French language,
* Absence of medical insurance,
* Participation in another intervention trial,
* Enforced hospitalization (ASPDT, ASPPI, ASPRE),
* Intellectuel Deficiency (IQ<70), and / or sensorimotor deficits incompatible with the cognitive training,

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary assessment criterion | Month 9
  The main outcome will be the global functioning measured by the Personal and Social Performance (PSP) Scale after 3 months of cognitive training . The PSP is a 100-point single-item rating scale. The ratings are done by a clinician, in 5-10 min, and require minimal training, with excellent inter-rater reliability. The scale considers four main areas:
  1. socially useful activities;
  2. personal and social relationships;
  3. self-care; and 4) disturbing and aggressive behaviours during a determined reference period (hereit will be the last month). It was found to be a quick and valid measure, sensitive to change, of patients; personal and social functioning even in early stage of psychosis.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Odile MO KREBS, PROFESSEUR, Principal Investigator — GHU PARIS Saint-Anne
Locations (1):
- Groupe Hospitalier Universitaire Paris - Psychiatrie et Neurosciences, (GHU Paris), Paris, France

IPD SHARING:
Plan to Share IPD: No